CLINICAL TRIAL: NCT01024842
Title: HIV-CORE 001 - A Randomised Placebo-controlled Study to Evaluate the Safety and Immunogenicity of a Candidate HIV-1 Vaccine, MVA.HIVconsv, Delivered by Intramuscular Needle Injection to HIV-1 Seropositive Adult Subjects Receiving Antiretroviral Therapy (ART).
Brief Title: Safety and Immunogenicity of MVA.HIVconsv in HIV-1 Seropositive Adults on HAART
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow recruitment therefore study was stopped after 95% volunteers were enrolled.
Sponsor: University of Oxford (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HIV-CORE 001
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: HIV-1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low dose vaccinees (Experimental): Individuals will receive three intramuscular injections of MVA.HIVconsv alone at a dose of 1x10^8 pfu.
  Interventions: Biological: MVA.HIVconsv low dose
- High dose vaccinees (Experimental): Individuals will receive three intramuscular injections of MVA.HIVconsv alone at a dose of 4x10^8 pfu.
  Interventions: Biological: MVA.HIVconsv high dose
- Low dose placebo (Placebo Comparator): Individuals will receive three intramuscular injections of low dose placebo
  Interventions: Other: Placebo low dose
- High dose placebo (Placebo Comparator): Individuals will receive three intramuscular injections of high dose placebo
  Interventions: Other: Placebo high dose

INTERVENTIONS:
Biological: MVA.HIVconsv low dose — Three intramuscular injections of MVA.HIVconsv alone at a dose of 1x10^8 pfu at week 0, 4 and 12.
  Arms: Low dose vaccinees
Other: Placebo low dose — Three intramuscular injections of placebo alone (200ul) at week 0, 4 and 12.
  Arms: Low dose placebo
Biological: MVA.HIVconsv high dose — Three intramuscular injections of MVA.HIVconsv alone at a dose of 4x10^8 pfu at week 0, 4 and 12.
  Arms: High dose vaccinees
Other: Placebo high dose — Three intramuscular injections of placebo alone (800ul) at week 0, 4 and 12.
  Arms: High dose placebo

SUMMARY:
In this study, the novel vaccine candidate, MVA.HIVconsv, will be tested for safety, tolerability and immunogenicity in HIV-1-seropositive subjects receiving effective antiretroviral therapy.

MVA.HIVconsv will be tested as a single vaccine modality, as a prelude to testing in a heterologous viral vector boost regimen which will include a replication-defective simian adenovirus expressing the same immunogen.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-60 years
* Confirmed HIV-1 seropositive
* Willing and able to give written informed consent for participation in the study
* Treated continuously with a combination of 3 or more antiretroviral agents for the preceding 12 months
* Willing and able to adhere to an effective ART regimen for the duration of the study (switching from current regimen is allowed if for reasons of tolerability or toxicity)
* CD4 cell count > 350 cells/μl at screening and at the preceding clinic visit
* Plasma viral load < 50 copies / ml at screening and at the preceding clinic visit
* No new AIDS-defining diagnosis or progression of HIV-related disease in the preceding 6/12 months
* Haematological and biochemical laboratory parameters as follows:

  * Haemoglobin > 10g/dl
  * Platelets > 100,000/μl
  * ALT ≤ 2.5 x ULN
  * Creatinine ≤ 1.3 x ULN
* Serology: negative for hepatitis B surface antigen OR HbsAg positive with HBV DNA < 1000 copies/ml; negative for hepatitis C antibodies OR confirmed clearance of HCV infection (spontaneous or following treatment); negative syphilis serology or documented adequate treatment of syphilis if positive EIA IgG or TPHA
* Available for follow up for duration of study (screening + 38 weeks) and willing to comply with the protocol requirements
* Women of child-bearing age must not be pregnant, planning a pregnancy or breast-feeding. Sexually active women must be willing to use an approved method of contraception from screening until 4 months after the third immunisation. Sexually active men in heterosexual relationships must be willing to use an approved method of contraception with their partners from screening until 4 months after the third immunisation.

Exclusion Criteria:

* Confirmed HIV-2 seropositive
* Positive pregnancy test
* Participation in another clinical trial within 12 weeks of study entry
* History of autoimmune disease other than HIV-related auto-immune disease which has resolved with ART
* History or clinical manifestations of any physical or psychiatric disorder which could impair the subject's ability to complete the study
* History of anaphylaxis or severe adverse reaction to vaccines
* History of alcohol or drug dependency which could, in the opinion of the investigators, impair the subject's ability to complete the study
* Previous immunisation with a recombinant MVA vaccine
* Immunisation with any experimental immunogens within 6 months of study entry
* Receipt of blood products or immunoglobulins within 6 months of study entry
* Treatment for cancer or lymphoproliferative disease within 1 year of study entry
* Receipt of vaccines other than Hepatitis B vaccine within 2 weeks of study entry or planned receipt within 2 weeks of vaccination
* Any other prior therapy which, in the opinion of the investigators, would make the individual unsuitable for the study or influence the results of the study
* Current or recent use (within last 3 months) of interferon or systemic corticosteroids or other immunosuppressive agents

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2009-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The proportion of volunteers who develop a grade 3 or 4 local or systemic reactions | Actively collected data throughout the study until 6 months after the last vaccination

SECONDARY OUTCOMES:
A descriptive summary of grade 3 or 4 local and systemic events, including laboratory abnormalities | Actively collected data throughout the study until 6 months after the last vaccination
A descriptive summary of serious adverse events, including laboratory abnormalities | Actively collected data throughout the study until 6 months after the last vaccination
The proportion of volunteers who develop CD8+ T cell responses to a new HIV-1 epitope, as determined by IFN-γ ELISPOT assay | Screen (≤ day -28); Day 0; Day 14; Day 28; Day 42; Day 56; Day 84; Day 112; Day 182; Final visit (day 266 / early termination)
The proportion of volunteers in whom the magnitude of CD8+ T cell responses to HIVconsv peptides increases by ≥ 3-fold, as determined by IFN-γ ELISPOT assay | Screen (≤ day -28); Day 0; Day 14; Day 28; Day 42; Day 56; Day 84; Day 112; Day 182; Final visit (day 266 / early termination)
Evaluation of the effect of MVA.HIVconsv vaccinations on viral suppressive capacity of CD8+ T cells in vitro, using a novel flow cytometric assay | Screen (≤ day -28); Day 0; Day 14; Day 28; Day 42; Day 56; Day 84; Day 112; Day 182; Final visit (day 266 / early termination)
Magnitude and phenotype, including but not limited to activation status, of HIV-1-specific CD8+ T cell populations identified by tetramer staining before and after vaccination, in selected volunteers with appropriate HLA class I alleles. | Screen (≤ day -28); Day 0; Day 14; Day 28; Day 42; Day 56; Day 84; Day 112; Day 182; Final visit (day 266 / early termination)
PBMC will be stored for other exploratory assays to characterise vaccine-expanded T cell populations such as IL-10 secretion and CFSE proliferation assays. | Screen (≤ day -28); Day 0; Day 14; Day 28; Day 42; Day 56; Day 84; Day 112; Day 182; Final visit (day 266 / early termination)
Serum and plasma will be stored for investigation of binding and neutralising antibodies to vaccinia and of pro-inflammatory cytokines. | Screen (≤ day -28); Day 0; Day 14; Day 28; Day 42; Day 56; Day 84; Day 112; Day 182; Final visit (day 266 / early termination)

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Hanke, Principal Investigator — University of Oxford; Andrew McMichael, Principal Investigator — University of Oxford; Lucy Dorrell, Principal Investigator — University of Oxford
Locations (2):
- United Kingdom (2):
  - Weatherall Institute of Molecular Medicine, Oxford, Oxons
  - Oxford Genitourinary Medicine, Oxford, Oxon

IPD SHARING:
Plan to Share IPD: Yes
Data are presented in a manuscript submitted to a peer-reviewed journal.

REFERENCES:
- [Derived] Hancock G, Moron-Lopez S, Kopycinski J, Puertas MC, Giannoulatou E, Rose A, Salgado M, Hayton EJ, Crook A, Morgan C, Angus B, Chen F, Yang H, Martinez-Picado J, Hanke T, Dorrell L. Evaluation of the immunogenicity and impact on the latent HIV-1 reservoir of a conserved region vaccine, MVA.HIVconsv, in antiretroviral therapy-treated subjects. J Int AIDS Soc. 2017 May 19;20(1):21171. doi: 10.7448/IAS.20.1.21171. PMID 28537062